CLINICAL TRIAL: NCT04960124
Title: An Open-Label, Parallel-Group, Single-Dose Study to Evaluate the Effect of Hepatic Impairment on the Pharmacokinetics, Safety, and Tolerability of JNJ-42847922 in Adult Participants
Brief Title: A Study to Evaluate the Effect of Hepatic Impairment on JNJ-42847922 in Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108929; 2020-005235-69 (EudraCT Number); 42847922MDD1012 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-07-02; First posted 2021-07-13 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy; Hepatic Impairment
MeSH Terms: interventions — seltorexant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1: Cohort 1 (JNJ-42847922) (Experimental): Participants with normal hepatic function will receive Dose 1 of JNJ-42847922 on Day 1.
  Interventions: Drug: JNJ-42847922
- Part 1: Cohort 2 (JNJ-42847922) (Experimental): Participants with mild hepatic impairment will receive Dose 1 of JNJ-42847922 on Day 1.
  Interventions: Drug: JNJ-42847922
- Part 1: Cohort 3 (JNJ-42847922) (Experimental): Participants with moderate hepatic impairment will receive Dose 2 of JNJ-42847922 on Day 1.
  Interventions: Drug: JNJ-42847922
- Part 2: Cohort 4 (Optional) (JNJ-42847922) (Experimental): Participants with moderate hepatic impairment will receive Dose 1 (depending on the results of Cohort 3) of JNJ-42847922 on Day 1.
  Interventions: Drug: JNJ-42847922
- Part 2: Cohort 5 (Optional) (JNJ-42847922) (Experimental): Participants with severe hepatic impairment will receive Dose 2 or Dose 3 (depending on the results of Part 1) of JNJ-42847922 on Day 1.
  Interventions: Drug: JNJ-42847922

INTERVENTIONS:
Drug: JNJ-42847922 — Participants will receive JNJ-42847922 tablet as a single oral dose (Dose 1 or Dose 2 or Dose 3) on Day 1.
  Other Names: Seltorexant

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (PK) of a single oral dose of JNJ-42847922 in adult participants with hepatic impairment when compared to healthy participants with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

All

* Be a man or woman 18 to 79 years of age, inclusive Participants with normal hepatic function
* Generally healthy
* Must not exceed upper limit of normal limits for serum bilirubin, transaminase levels, albumin levels, prothrombin time (PT), and International Normalized Ratio (INR) when measured at screening and Day 1 Participants with (Mild, Moderate or Severe) hepatic impairment
* Medically stable
* Total Child-Pugh score of 5 or 6, inclusive (mild); or 7 to 9, inclusive (moderate); or 10 to 15, inclusive (severe) as determined by the investigator
* Stable hepatic function during screening and those measured on Day 1
* Stable renal function

Exclusion Criteria:

Participants with normal hepatic function

* Hepatitis B surface antigen (HBsAg) or hepatitis C antibodies at screening Participants with (Mild, Moderate or Severe) hepatic impairment
* Severe ascites or pleural effusion; prothrombin time greater than (>)18 seconds; evidence of progressive liver disease within the previous 4 weeks, as indicated by changes in hepatic transaminases, alkaline phosphatase, and gamma-glutamyl transferase
* History of hepatopulmonary syndrome, hydrothorax, or significant hepatorenal syndrome
* Acute or exacerbating hepatitis, fluctuating or rapidly deteriorating hepatic function as indicated by widely varying or worsening of clinical and/or laboratory signs of hepatic impairment in the judgment of either the investigator or the sponsor's medical monitor
* Clinically significant laboratory findings except as related to hepatic impairment

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2021-11-19 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Analyte Concentration (Cmax) of JNJ-42847922 and its Metabolites M12 and M16 | Pre-dose, up to 96 hours post-dose (up to Day 5)
  Cmax is defined as maximum observed plasma analyte concentration of JNJ-42847922 and its metabolites M12 and M16.
Area Under Plasma Analyte Concentration versus Time Curve from Time Zero to Time of Last Measurable Concentration (AUC [0-last]) of JNJ-42847922 and its Metabolites M12 and M16 | Pre-dose, up to 96 hours post-dose (up to Day 5)
  AUC(0-last) is defined as area under the plasma analyte concentration versus time curve from time zero to time of last measurable concentration of JNJ-42847922 and its metabolites M12 and M16.
Area Under the Plasma Analyte Concentration versus Time Curve from Time Zero to Infinite Time (AUC[0-Infinity]) of JNJ-42847922 and its Metabolites M12 and M16 | Pre-dose, up to 96 hours post-dose (up to Day 5)
  AUC(0-infinity) is defined as the area under the plasma analyte concentration versus time curve from time zero to infinite time of JNJ-42847922 and its metabolites M12 and M16.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Up to Day 5
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (2):
- Germany (2):
  - CRS Clinical Research Services Kiel GmbH, Kiel
  - APEX GmbH, München

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson and Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency